CLINICAL TRIAL: NCT03284684
Title: Kinetics of Perioperative Circulating DNA in Cancer Surgery
Acronym: Periop ctDNA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016/PC-01; 2017-A00950-53 (Other: ANSM)
Record Dates: First submitted 2017-08-08; First posted 2017-09-15 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Prostate Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- circulating DNA plasma level test
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — plasma concentration of circulating DNA of specific genes

SUMMARY:
The aim of this study was to determine the kinetics of perioperative circulating DNA in three types of cancer. This first step will enable further studies comparing the potential impact of certain techniques or anesthetic products on cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is aged between 18-75
* Patient must weigh >40kg
* The patient will receive adjusted carcinological surgery
* Indication of curative surgery
* The patient has already undergone tumoral biopsy prior to surgery
* The patient has stage M0 cancer of either colon (right or left colonic adenocarcinoma), prostate (adenocarcinoma) or breast (infiltrating carcinoma)

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is pregnant, parturient or breast feeding
* Chronic alcoholism
* The patient has received radiotherapy or chemotherapy periopratively
* Cancer other than colon, breast or prostate
* The patient has currently or in the past, had a cancerous lesion
* Neo-adjuvant therapy (immunotherapy, radiotherapy, chemotherapy)
* Emergency cancer surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for non-metastatic solid tumors: colon, breast and prostate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Change in concentration of total mutant circulating DNA | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in proportion of mutant circulating DNA | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in integrity index of circulating DNA for ACTB gene | Nine timepoints between Day-1 to Day 3
  concentration of long ACTB ctDNA fragments/concentration of short ACTB ctDNA fragments
Change in integrity index of circulating DNA for KRAS gene | Nine timepoints between Day-1 to Day 3
  concentration of long KRAS ctDNA fragments/concentration of short KRAS ctDNA fragments

SECONDARY OUTCOMES:
Change in plasma concentration of long (~ 290bp) fragments of ACTB gene | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in plasma concentration of short (~ 145bp) fragments of KRAS gene | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in plasma concentration of long (~ 300bp) fragments of KRAS gene | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in plasma concentration of mutant KRAS DNA fragments | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma
Change in plasma concentration of BRAF DNA fragments with V600E mutation | Nine timepoints between Day-1 to Day 3
  ng/mL in plasma

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Montpellier, Montpellier
  - Institut de Cancérologie Montpellier, Montpellier
  - CHU Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kudriavtsev A, Pastor B, Mirandola A, Pisareva E, Gricourt Y, Capdevila X, Thierry AR, Cuvillon P. Association of the immediate perioperative dynamics of circulating DNA levels and neutrophil extracellular traps formation in cancer patients. Precis Clin Med. 2024 Mar 27;7(2):pbae008. doi: 10.1093/pcmedi/pbae008. eCollection 2024 Jun. PMID 38699382